CLINICAL TRIAL: NCT03002311
Title: Improving Medical Care With Electronic Interventions Based on Automated Text and Phone Messages
Brief Title: Improving Follow-Up for Discharged Emergency Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Epharmix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201504079
Record Dates: First submitted 2016-11-23; First posted 2016-12-23 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: General Medicine; Emergency Medicine; Mobile Health
Keywords: Bioinformatics; Electronic pharmacology; Mobile health; Electronic health; Adherence; Digital health; Health information technology; mHealth; eHealth

STUDY DESIGN:
Intervention Model Description: SMS text messaging to prompt adherence with follow-up appointment.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Receiving current standard of care as designated by emergency department (ED) standard operating practice.
- Epharmix/CareSignal eHealth Intervention (Experimental): After randomization, participants receive text reminders to have a follow-up visit. The participant can respond to these messages via numerical or binary answers (Y/N).
  Interventions: Device: Epharmix/CareSignal eHealth

INTERVENTIONS:
Device: Epharmix/CareSignal eHealth — The self-scheduling text and phone messaging system was built by Epharmix/CareSignal. Participants in the intervention group began receiving text or voice messages (for landlines) starting 1 hour following ED discharge if during normal business hours, or at 1000 the next business morning. Automated messages were sent up to 3 days in a row or until the participant responded or opted out. The phone system would ultimately connect them directly to their referral provider or clinic to schedule an appointment. Once participants hung up with the referral clinic, the intervention texted or called back to solicit the appointment date. If a date was entered, the system sent reminders at 14 days, 7 days, 3 days, and 1 day before the appointment. After the appointment, the intervention texted or called participants to confirm if they attended.
  Arms: Epharmix/CareSignal eHealth Intervention

SUMMARY:
This study's purpose is to test the effects of an electronic health intervention platform developed by Epharmix (also known as CareSignal), which features two-way SMS text messages and phone calls intended to improve clinical outcomes compared to the standard of care. This was a randomized open, blinded end-point (PROBE) trial of adult patients discharged from the ED and referred to a provider for follow-up care. Participants in the intervention arm received a self-scheduling text or phone message that automatically connected them to their referral provider to schedule a follow-up appointment and sent them appointment reminders. Those in the control arm received standard of care written instructions to contact listed referral providers. The primary outcome was time to the follow-up appointment.

DETAILED DESCRIPTION:
Telemedicine is a modern field of clinical medicine that strives to incorporate telecommunication and information technology for diagnosing and managing health care at a distance. Interventions range from telephone reminders to remote physician consultation by streamed by webcam. Simple technology such as telephone and SMS texting are becoming common forms of communication and may improve patient adherence and engagement. Automated telephone appointment reminders have improved adherence with follow-up appointments in some settings, but have mixed results in patients discharged from the emergency department (ED). Increasing adherence to follow-up care has been a priority in the ED to improve patient outcomes and reduce unnecessary future visits.

An electronic intervention platform has been developed by Epharmix (now HealthSignal), uses SMS text messaging for adherence tracking and data collection applications, to supplement clinical care. Specific messages include: proactively asking patients or a designated patient advocate if the patient has experienced a medical event; requesting specific care-related information; and providing health care education. Patients receiving the messages are also provided with key contact information for their designated health care provider to promote patient engagement, as well as prompt and appropriate medical follow-up care. The service will maintain both a dedicated SMS and phone line for recording events or adverse reactions. Events designated as critical prompt a phone call from nursing staff. Overall, this study aims to determine whether an electronic intervention system that sends SMS text messages will improve adherence to follow-up appointments after an ED visit.

Patients age 18 years or older at Barnes Jewish Hospital are included in this study. We conducted a prospective randomized open, blinded end-point (PROBE) trial of 278 adult patients discharged from the ED and referred to a provider for follow-up care. Participants in the intervention arm received a self-scheduling text or phone message using the Epharmix (now HealthSignal) platform that connected them to their referral provider to schedule a follow-up appointment and sent them appointment reminders. Those in the control arm received standard-of-care written instructions to contact listed referral providers. The primary outcome was time to appointment. The secondary outcome was time to return visit to the ED.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older,
2. accessible short message service (SMS) capable mobile phone or residential landline,
3. able to read English or have English-speaking family member to assist with phone communications,
4. discharged directly from the Barnes Jewish hospital (St. Louis, MO) emergency department (ED), and
5. given a clinical referral to make an outpatient follow-up appointment at time of discharge to a specific clinic or provider

Exclusion Criteria:

1. unable or refused to provide consent,
2. could not be contacted by a phone call or SMS,
3. non-English speaking,
4. were admitted to the hospital, and
5. already had a follow-up appointment scheduled before being discharged from the ED

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Will R Ross, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes Jewish Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Whittier WL. Surveillance of hemodialysis vascular access. Semin Intervent Radiol. 2009 Jun;26(2):130-8. doi: 10.1055/s-0029-1222457. PMID 21326504
- [Background] Cummings KM, Becker MH, Kirscht JP, Levin NW. Intervention strategies to improve compliance with medical regimens by ambulatory hemodialysis patients. J Behav Med. 1981 Mar;4(1):111-27. doi: 10.1007/BF00844851. PMID 7288877
- [Background] Parikh A, Gupta K, Wilson AC, Fields K, Cosgrove NM, Kostis JB. The effectiveness of outpatient appointment reminder systems in reducing no-show rates. Am J Med. 2010 Jun;123(6):542-8. doi: 10.1016/j.amjmed.2009.11.022. PMID 20569761
- [Background] Junod Perron N, Dao MD, Righini NC, Humair JP, Broers B, Narring F, Haller DM, Gaspoz JM. Text-messaging versus telephone reminders to reduce missed appointments in an academic primary care clinic: a randomized controlled trial. BMC Health Serv Res. 2013 Apr 4;13:125. doi: 10.1186/1472-6963-13-125. PMID 23557331
- [Background] Bame SI, Petersen N, Wray NP. Variation in hemodialysis patient compliance according to demographic characteristics. Soc Sci Med. 1993 Oct;37(8):1035-43. doi: 10.1016/0277-9536(93)90438-a. PMID 8235736
- [Background] Lua PL, Neni WS. A randomised controlled trial of an SMS-based mobile epilepsy education system. J Telemed Telecare. 2013 Jan;19(1):23-8. doi: 10.1177/1357633X12473920. Epub 2013 Feb 6. PMID 23390210
- [Background] Lua PL, Neni WS. Health-related quality of life improvement via telemedicine for epilepsy: printed versus SMS-based education intervention. Qual Life Res. 2013 Oct;22(8):2123-32. doi: 10.1007/s11136-013-0352-6. Epub 2013 Jan 18. PMID 23329469
- [Background] Dall TM, Storm MV, Chakrabarti R, Drogan O, Keran CM, Donofrio PD, Henderson VW, Kaminski HJ, Stevens JC, Vidic TR. Supply and demand analysis of the current and future US neurology workforce. Neurology. 2013 Jul 30;81(5):470-8. doi: 10.1212/WNL.0b013e318294b1cf. Epub 2013 Apr 17. PMID 23596071
- [Background] Lieberman DZ, Kelly TF, Douglas L, Goodwin FK. A randomized comparison of online and paper mood charts for people with bipolar disorder. J Affect Disord. 2010 Jul;124(1-2):85-9. doi: 10.1016/j.jad.2009.10.019. Epub 2009 Nov 6. PMID 19896202
- [Background] Sawan M, Salam MT, Le Lan J, Kassab A, Gelinas S, Vannasing P, Lesage F, Lassonde M, Nguyen DK. Wireless recording systems: from noninvasive EEG-NIRS to invasive EEG devices. IEEE Trans Biomed Circuits Syst. 2013 Apr;7(2):186-95. doi: 10.1109/TBCAS.2013.2255595. PMID 23853301
- [Background] Chaudhry SI, Mattera JA, Curtis JP, Spertus JA, Herrin J, Lin Z, Phillips CO, Hodshon BV, Cooper LS, Krumholz HM. Telemonitoring in patients with heart failure. N Engl J Med. 2010 Dec 9;363(24):2301-9. doi: 10.1056/NEJMoa1010029. Epub 2010 Nov 16. PMID 21080835
- [Result] Bauer KL, Sogade OO, Gage BF, Ruoff B, Lewis L. Improving Follow-up Attendance for Discharged Emergency Care Patients Using Automated Phone System to Self-schedule: A Randomized Controlled Trial. Acad Emerg Med. 2021 Feb;28(2):197-205. doi: 10.1111/acem.14080. Epub 2020 Aug 5. PMID 32654257
- [Derived] Chen RY, Feltes JR, Tzeng WS, Lu ZY, Pan M, Zhao N, Talkin R, Javaherian K, Glowinski A, Ross W. Phone-Based Interventions in Adolescent Psychiatry: A Perspective and Proof of Concept Pilot Study With a Focus on Depression and Autism. JMIR Res Protoc. 2017 Jun 16;6(6):e114. doi: 10.2196/resprot.7245. PMID 28623183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period for the study took place between January 1, 2016 and June 30, 2017.
Pre-assignment Details: Of 933 patients screened, 35% were enrolled. Of those screened, 4.5% of patients were excluded because they did not have a phone and 2.0% were excluded because they were non-English speaking. The largest groups excluded were those who did not want to participate (n=300) and those who were given a specific referral (n=107).
Groups:
- Epharmix/CareSignal eHealth Intervention: Epharmix/CareSignal eHealth: The self-scheduling text and phone messaging system was built by Epharmix/CareSignal. Participants in the intervention group began receiving text or voice messages (for landlines) starting 1 hour following ED discharge if during normal business hours, or at 1000 the next business morning. Automated messages were sent up to 3 days in a row or until the participant responded or opted out. The phone system would ultimately connect them directly to their referral provider or clinic to schedule an appointment. Once participants hung up with the referral clinic, the intervention texted or called back to solicit the appointment date. If a date was entered, the system sent reminders at 14 days, 7 days, 3 days, and 1 day before the appointment. After the appointment, the intervention texted or called participants to confirm attendance.
Period: Overall Study
Arm/Group | Control | Epharmix/CareSignal eHealth Intervention
Started | 147 | 180
Completed | 128 | 150
Not Completed | 19 | 30
Not completed — Lost to Follow-up | 13 | 26
Not completed — Referral provider called to schedule app | 3 | 3
Not completed — Physician Decision | 3 | 1

BASELINE CHARACTERISTICS:
Population: 19 patients in the control arm were excluded: 3 were admitted to the hospital, 3 had their provider schedule an appointment, and 13 had no outcome data.
  30 patients in the phone intervention arm were excluded: 1 was admitted to the hospital, 3 had their provider schedule an appointment, and 26 had no outcome data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Epharmix/CareSignal eHealth Intervention | Total
Number analyzed (Participants) | 128 | 150 | 278
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36.5 [26.5 to 48.0] | 38.4 [27.3 to 54.3] | 37.5 [27 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 98 | 180
  Male | 46 | 52 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 5 | 8
  Not Hispanic or Latino | 124 | 143 | 267
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 87 | 100 | 187
  White | 30 | 40 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 128 | 150 | 278

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Follow-up Appointment
Description: The primary outcome was the effect of the intervention on time to follow-up appointment using an intention-to-treat analysis and plotting the cumulative incidence functions (CIFs). Follow-up adherence was defined as a recorded visit in the EMR to the referral primary or specialty care provider within 120 days after ED discharge to address a similar diagnosis (or complaint) at the index ED visit.
Time Frame: Up to 120 days
Population: Modified intent-to treat-analysis: Participants were excluded if they were admitted to the hospital after consenting, if their doctor called to schedule the follow-up appointment, or if they were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Epharmix/CareSignal eHealth Intervention
Number analyzed (Participants) | 128 | 150
Participants | 30 | 74
Statistical Analysis 1: Comparison: Control vs Epharmix/CareSignal eHealth Intervention; Test type: Superiority — We conducted a conditional power analysis 120 days after 6 months of enrollment. We determined the effect size based on the difference of proportions of follow-up attendance in the intervention and control arms. We used the effect size of 20% to estimate the sample size needed for a two-sided alpha of 0.05 at 90% power and a 1:1 ratio to require 266 participants. Loss to follow-up was estimated to be 20%, increasing target enrollment to 334 total participants; p < 0.001, Gray's test; We compared the cumulative incidence function

2. Secondary Outcome: Revisits to the ED
Description: The secondary outcome was revisits to the ED after discharge.
Time Frame: Up to 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Epharmix/CareSignal eHealth Intervention
Number analyzed (Participants) | 128 | 150
Participants | 50 | 60
Statistical Analysis 1: Comparison: Control vs Epharmix/CareSignal eHealth Intervention; Test type: Superiority — This was a secondary analysis so no power analysis was done; p = 0.8, Gray's test — We used a two-sided alpha of 0.05 to determine significance; We compared the cumulative incidence functions

ADVERSE EVENTS:
Time Frame: 120 days
Description: SAEs consisted of deaths (none observed) or unplanned hospital admissions (see table).
Arm/Group | Control | Epharmix/CareSignal eHealth Intervention
All-Cause Mortality (participants affected / at risk) | 0/128 | 0/150
Serious Adverse Events (participants affected / at risk) | 16/128 | 16/150
Other Adverse Events (participants affected / at risk) | 0/128 | 0/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=128) | Epharmix/CareSignal eHealth Intervention (N=150)
Unplanned hospitalization (General disorders) | 16 (16) | 16 (16) — Unplanned hospitalizations consisted of non-elective hospitalizations within the 120-day windom.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT03002311/Prot_SAP_ICF_000.pdf